CLINICAL TRIAL: NCT06728046
Title: Analgesic Effects of Ultrasound-Guided Erector Spinae Plane Block v.s Patient Controlled Analgesia in Correction Surgery for Idiopathic Scoliosis: A Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block v.s Patient Controlled Analgesia in Correction Surgery for Idiopathic Scoliosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCH20241202
Record Dates: First submitted 2024-12-01; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Scoliosis; Erector Spinae Plane Block; Patient Controlled Analgesia
Keywords: Erector Spinae Plane Block; Patient Controlled Analgesia; Idiopathic Scoliosis Correction Surgery
MeSH Terms: interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to differences in clinical management between the groups, investigators, participants, and clinical staff will be aware of group assignments. However, follow-up researchers and statisticians responsible for data analysis will remain blinded to the group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB Group (Experimental): Participants will receive ultrasound-guided ESPB preoperatively, using 40 ml of 0.3% ropivacaine.
  Interventions: Other: ESPB
- PCA Group (Active Comparator): Participants will receive postoperative PCA with a formulation of 200 µg sufentanil diluted to 100 ml. The PCA settings will include a background dose of 3 ml/hour, a lockout time of 15 minutes, and a bolus dose of 2 ml.
  Interventions: Device: PCA

INTERVENTIONS:
Other: ESPB — Participants will receive ultrasound-guided ESPB preoperatively, using 40 ml of 0.3% ropivacaine.
  Arms: ESPB Group
Device: PCA — Participants will receive postoperative PCA with a formulation of 200 µg sufentanil diluted to 100 ml. The PCA settings will include a background dose of 3 ml/hour, a lockout time of 15 minutes, and a bolus dose of 2 ml.
  Arms: PCA Group

SUMMARY:
Scoliosis correction surgery involves extensive surgical wounds, intense intraoperative stimulation, and severe postoperative pain, often necessitating the use of potent opioids. However, there is a critical clinical need for effective pain management strategies that both ensure sufficient analgesia and minimize opioid-related adverse effects. The Erector Spinae Plane Block (ESPB) has shown promise as an effective analgesic technique, but its application in scoliosis correction surgery has not been reported.We hypothesize that ESPB provides superior postoperative analgesia compared to patient-controlled intravenous analgesia (PCA) pumps. Specifically, ESPB is expected to significantly reduce postoperative pain scores, decrease perioperative opioid consumption, and mitigate opioid-related side effects.

This study is a randomized controlled trial involving 40 participants undergoing scoliosis correction surgery, randomized into two groups: the ESPB group and the PCA group. The primary outcome measure is the resting pain score at 2 hours postoperatively, which will be used to evaluate the efficacy of ESPB. Secondary outcomes include perioperative opioid consumption and the incidence of opioid-related adverse effects. The study aims to provide evidence for ESPB as an innovative and effective method for postoperative analgesia in scoliosis correction surgery.

DETAILED DESCRIPTION:
Scoliosis correction surgery involves large surgical wounds spanning multiple vertebrae, requiring sufficient analgesia to manage intense intraoperative stimulation and severe postoperative pain. Effective pain control in this context often necessitates potent opioids, such as morphine or equivalent drugs. Current perioperative analgesia strategies include intraoperative use of long-acting opioids (e.g., sufentanil, fentanyl) and patient-controlled analgesia (PCA) pumps for postoperative pain management, primarily involving opioids like sufentanil or morphine. However, opioids are associated with adverse effects such as nausea, vomiting, bowel obstruction, pruritus, dizziness, respiratory depression, opioid tolerance, and hyperalgesia, which can lead to suboptimal pain control and negatively impact patients' quality of life and postoperative recovery. There is a critical need for effective analgesic methods in scoliosis correction surgery that minimize opioid-related adverse effects, enhance the patient experience, and promote accelerated recovery.

The Erector Spinae Plane Block (ESPB) was first reported by Forero et al. in 2016 as an effective analgesic technique for rib-related neuropathic pain. Its mechanism involves the injection of local anesthetics into the fascial plane between the erector spinae muscle and the transverse process, allowing for the diffusion of the anesthetic to adjacent areas. ESPB exerts its primary analgesic effect through the posterior branches of spinal nerves and can further diffuse anteriorly to paravertebral and epidural spaces, and laterally across the costotransverse foramina, affecting nerve roots and visceral structures. This mechanism provides comprehensive analgesia. ESPB has since been widely applied in perioperative pain management for thoracic surgery, shoulder arthroscopy, breast surgery, abdominal surgery, cesarean sections, and urological procedures, as well as for acute and chronic pain conditions such as rib fractures, postherpetic neuralgia, burns, and cancer pain.

Studies have demonstrated that ESPB effectively reduces postoperative pain scores, decreases opioid consumption, delays the need for rescue analgesics, reduces the number of patients requiring rescue medication, and lowers the incidence of nausea and vomiting in spinal surgeries. Although there are limited case reports and clinical experience summarizing its perioperative analgesic effect in scoliosis correction surgery, preliminary findings suggest it is effective.

Based on the analgesic mechanism of ESPB and prior studies, we hypothesize that ESPB provides superior postoperative pain control compared to PCA, significantly reducing postoperative pain scores, perioperative opioid consumption, and associated adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 years or older, regardless of gender.
* Scheduled for scoliosis correction surgery.
* Signed informed consent from the participant or their legal guardian.

Exclusion Criteria:

* Allergy to local anesthetics such as ropivacaine.
* Family history of malignant hyperthermia.
* Severe systemic diseases affecting the heart, lungs, liver, or kidneys.
* Neurological or psychiatric disorders.
* Communication difficulties, such as hearing impairment or speech disorders.
* Concurrent participation in other clinical studies.
* Other conditions deemed unsuitable for participation by the investigators.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Resting numerical rating scale (NRS) pain scores | 2 hours postoperatively
  The Numerical Rating Scale (NRS) is a tool for assessing pain intensity, allowing patients to rate their pain on a scale from 0 to 10, where 0 represents "no pain," 10 represents "the worst pain imaginable," and pain levels are categorized as 0 (no pain), 1-3 (mild pain), 4-6 (moderate pain), and 7-10 (severe pain).

SECONDARY OUTCOMES:
Severe complications | 30 days postoperatively
  The incidence of severe complications are categorized into five grades based on severity: Grade I (resolved with temporary treatment, e.g., postoperative nausea and vomiting), Grade II (prolonged hospital stay required, e.g., pneumonia requiring antibiotics), Grade III (life-threatening events requiring intervention but recoverable during hospitalization, e.g., deep vein thrombosis), Grade IV (significant harm persisting 30 days or longer with a marked decrease in quality of life, e.g., postoperative cognitive dysfunction or delirium), and Grade V (death within 30 days postoperatively).
Postoperative resting NRS pain scores | 3 days after surgery
  Resting NRS pain scores on postoperative days 1, 2, and 3
Postoperative NRS pain scores during movement | 3 days after surgery
  NRS pain scores during movement on postoperative days 1, 2, and 3.
Postoperative opioids consumption | 30 days postoperatively
  Opioids will be used as a rescue measure for acute pain, including sulfentanil, fentanil, and morphine. Sulfentanil or fentanil will be given to the participants in PACU when the NRS scores higher than 4. When a participant's resting NRS pain score exceeds 4 in the ward, 5 mg of morphine can be administered intravenously. If the effect is insufficient, an additional 5 mg may be given after 30 minutes, with a maximum daily dose of 20 mg.
Time to initiate functional exercises | 30 days postoperatively
  Duration from hospital admission to the first attempt at mobilization, either preoperatively or postoperatively (in days)
Total length of hospital stay | 7 days after discharge
  Duration from hospital admission to discharge (in days)
Postoperative length of hospital stay | 7 days after discharge
  Duration from the day of surgery to discharge (in days)
Total hospital cost | 7 days after discharge
  Total hospital cost

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared after de-identification.The shared data will include de-identified individual participant data, and metadata supporting the primary and secondary outcomes, as well as the study protocol.Data will be available beginning 6 months after publication of the main study results and ending 3 years following publication. Requests for data sharing should be directed to the corresponding author (liaoren7733@163.com). Upon approval of a formal proposal, a data-sharing agreement will be signed, and access will be granted through a secure datasharing platform.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months after publication of the main study results and ending 3 years following publication.
Access Criteria: Requests for data sharing should be directed to the corresponding author: liaoren7733@163.com.

REFERENCES:
- [Derived] Liao C, Zhong J, Lai X, Liao R. Analgesic effects of bilateral ultrasound-guided erector spinae plane block versus patient controlled intravenous analgesia in correction surgery for idiopathic scoliosis: study protocol for a randomized controlled trial. Perioper Med (Lond). 2025 Nov 14;14(1):127. doi: 10.1186/s13741-025-00622-9. PMID 41239513